CLINICAL TRIAL: NCT02576535
Title: Protocol for Staged Stereotactic Radiosurgery for Large Arteriovenous Malformations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8844
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Intracranial Arteriovenous Malformations (AVM)
MeSH Terms: conditions — Intracranial Arteriovenous Malformations | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fractionated stereotactic radiosurgery (Experimental): The radiation dose will be delivered by the standard, FDA approved Leksell gamma unit (Gamma knife; Elekta Instruments, Atlanta, GA). Treatment dose and volume will be determined using the Gamma Plan software provided with the unit (Elekta Instruments, Atlanta, GA).
  Interventions: Procedure: Fractionated stereotactic radiosurgery; Device: Leskell gamma unit

INTERVENTIONS:
Procedure: Fractionated stereotactic radiosurgery
Device: Leskell gamma unit — FDA approved device
  Other Names: Gamma Knife

SUMMARY:
Stereotactic radiosurgery is a well established treatment option for arteriovenous malformations (AVMs). The potential complications related to radiosurgery are well documented and are predominately related to radiation effects to the surrounding brain parenchyma. These risks increase with larger lesions, requiring a concommitant reduction in the amount of radiation that can be delivered. This reduction in radiation dose decreases the efficacy of treatment. The broad, long-term objectives of this proposal are 1) to determine the role of fractionated stereotactic radiosurgery in the treatment of large (>10cc) AVMs; 2) to evaluate the complication rates related to fractionating these doses compared to conventional stereotactic treatment 3) to evaluate the success rate of treating large AVMs with this protocol.

DETAILED DESCRIPTION:
This research project will involve performing a preoperative MRI and angiogram on patients harboring an AVM to determine the feasibility of treating the lesion with gamma knife radiosurgery. Patient with lesions greater than 10 cc will be studied.

Each patient will have a Magnetic resonance angiography (MRA) with gadolinium and an angiogram immediately before each radiation treatment. If there is a contraindication for MRI examination (pacemaker or any other implanted ferromagnetic material), a CT angiogram will be obtained instead. Each treatment will be spaced at least 3 months apart. Follow-up MRIs or CT scans will be obtained at 6 month intervals. A follow-up angiogram will be obtained when there is radiographic evidence of complete occlusion based on the MRI images, or at 3 years after the procedure, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 or older
* Inpatients and outpatients, referred for radiosurgical treatment of an arteriovenous malformation
* Patients with lesions greater than 10 cc, who are currently symptomatic from the AVM (hemorrhage, seizure, or ischemia from steal phenomenon)

Exclusion Criteria:

* Patients without symptoms related to AVM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2000-02; Primary Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Huang, MD, Principal Investigator — NYU Langone Medical Center

RESULTS

PARTICIPANT FLOW:
Groups:
- Fractionated Stereotactic Radiosurgery: The radiation dose will be delivered by the standard, FDA approved Leksell gamma unit (Gamma knife; Elekta Instruments, Atlanta, GA). Treatment dose and volume will be determined using the Gamma Plan software provided with the unit (Elekta Instruments, Atlanta, GA).
  Fractionated stereotactic radiosurgery
  Leskell gamma unit: FDA approved device
Period: Overall Study
Arm/Group | Fractionated Stereotactic Radiosurgery
Started | 18
Completed | 16
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 16
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Asian or Pacific Islander | 3
  Black, not of Hispanic-American Origin | 4
  Hispanic-American | 4
  White, not of Hispanic-American Origin | 7
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Presence of T2 Weighted Changes on Serial MRI Exam Not Associated With Neurological Symptoms
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 16
participants | 3

2. Primary Outcome: Number of Participants With Presence of T2 Weighted Changes on Serial MRI Exam Associated With New Neurological Symptoms
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 16
participants | 2

3. Primary Outcome: Number of Participants With Presence of New Neurological Symptoms Without Evidence of MRI Abnormalities
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 16
participants | 2

4. Primary Outcome: Number of Participants Experiencing Hemorrhage From the Arteriovenous Malformation (AVM)
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 16
participants | 4

5. Primary Outcome: Number of Participants With Complete Occlusion of AVM on Serial MRI Confirmed With Angiography
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 16
participants | 15

6. Post Hoc Outcome: Number of Participants Experiencing Seizures
Time Frame: 10 years
Measure: Number; unit: participants
Arm/Group | Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 16
participants | 3

ADVERSE EVENTS:
Arm/Group | Fractionated Stereotactic Radiosurgery
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes